CLINICAL TRIAL: NCT02149186
Title: Interactive Motor Imagery in Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK-24 2009/PB_2016-00545
Record Dates: First submitted 2014-04-24; First posted 2014-05-29 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Spinal Cord Injury; Stroke
MeSH Terms: conditions — Spinal Cord Injuries; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rehabilitation (Experimental)
  Interventions: Device: iCTuS-L

INTERVENTIONS:
Device: iCTuS-L

SUMMARY:
This project will build and test the first rehabilitation system employing virtual reality (VR)-based observation, motor imagery and execution to treat lower-limb neuropathic pain and motor dysfunction in participants with an incomplete spinal cord injury or another neurological disorder, eg. stroke: iCTuS-L (Interactive Computer-based Therapy System for legs). Patients using the system will control virtual representations of their legs to engage in entertaining gaming interactions.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 and 80
* clinically incomplete spinal cord injury (time since injury: chronic > 1 year; acute < 3 months)
* ASI C or D
* neuropathic pain and/or motor deficits
* diagnosed neurological disorder, eg. stroke

Exclusion Criteria:

* any disease limiting training
* epilepsy
* major depression or psychosis

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sensorimotor Assessment | 16 weeks
  Questionnaire assessing distinct pain qualities associated with neuropathic pain, structured pain interview, questionnaire for assessing patients diagnosed as depressed and detects depression among the normal population, transcutaneous electrical stimulation of superficial nerves, information about the motor level of the lesion, the sensory levels of the lesion (light touch and pin prick), questionnaire assessing activities of daily life and independence in subjects with spinal cord lesion, walking aids and/or personal assistance, examining gait speed, transcranial magnetic stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Curt, Armin, MD, Zurich, Switzerland

REFERENCES:
- [Derived] Villiger M, Liviero J, Awai L, Stoop R, Pyk P, Clijsen R, Curt A, Eng K, Bolliger M. Home-Based Virtual Reality-Augmented Training Improves Lower Limb Muscle Strength, Balance, and Functional Mobility following Chronic Incomplete Spinal Cord Injury. Front Neurol. 2017 Nov 28;8:635. doi: 10.3389/fneur.2017.00635. eCollection 2017. PMID 29234302